CLINICAL TRIAL: NCT02601937
Title: A Phase 1 Study of the EZH2 Inhibitor Tazemetostat in Pediatric Subjects With Relapsed or Refractory INI1-Negative Tumors or Synovial Sarcoma
Brief Title: EZH2 Inhibitor Tazemetostat in Pediatric Subjects With Relapsed or Refractory INI1-Negative Tumors or Synovial Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EZH-102; 2015-002468-18 (EudraCT Number)
Record Dates: First submitted 2015-10-21; First posted 2015-11-11 (Estimated); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-06

CONDITIONS: Rhabdoid Tumors; INI1-negative Tumors; Synovial Sarcoma; Malignant Rhabdoid Tumor of Ovary
MeSH Terms: conditions — Rhabdoid Tumor; Sarcoma, Synovial | interventions — tazemetostat

STUDY DESIGN:
Intervention Model Description: Participants were enrolled either to the dose escalation or the dose expansion portion of the study. Participants in the dose expansion portion of the study were separated into cohorts based on their disease-type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Dose Escalation Level 1 (Experimental): Pediatric patients with select R/R rhabdoid tumors, INI1- SMARCA4-negative tumors, or synovial sarcoma who participated in the dose escalation portion of the study.
  Participants received 240 mg/m^2, open-label, oral tazemetostat twice daily (BID) in continuous 28-day cycles
  Interventions: Drug: Tazemetostat
- Dose Escalation Level 2 (Experimental): Pediatric patients with select R/R rhabdoid tumors, INI1- SMARCA4-negative tumors, or synovial sarcoma who participated in the dose escalation portion of the study.
  Participants received 300 mg/m^2, open-label, oral tazemetostat twice daily (BID) in continuous 28-day cycles
  Interventions: Drug: Tazemetostat
- Dose Escalation Level 3 (Experimental): Pediatric patients with select R/R rhabdoid tumors, INI1- SMARCA4-negative tumors, or synovial sarcoma who participated in the dose escalation portion of the study.
  Participants received 400 mg/m^2, open-label, oral tazemetostat twice daily (BID) in continuous 28-day cycles
  Interventions: Drug: Tazemetostat
- Dose Escalation Level 4 (Experimental): Pediatric patients with select R/R rhabdoid tumors, INI1- SMARCA4-negative tumors, or synovial sarcoma who participated in the dose escalation portion of the study.
  Participants received 520 mg/m^2, open-label, oral tazemetostat twice daily (BID) in continuous 28-day cycles
  Interventions: Drug: Tazemetostat
- Dose Escalation Level 5 (Experimental): Pediatric patients with select R/R rhabdoid tumors, INI1- SMARCA4-negative tumors, or synovial sarcoma who participated in the dose escalation portion of the study.
  Participants received 700 mg/m^2, open-label, oral tazemetostat twice daily (BID) in continuous 28-day cycles
  Interventions: Drug: Tazemetostat
- Dose Escalation Level 6 (Experimental): Pediatric patients with select R/R rhabdoid tumors, INI1- SMARCA4-negative tumors, or synovial sarcoma who participated in the dose escalation portion of the study.
  Participants received 900 mg/m^2, open-label, oral tazemetostat twice daily (BID) in continuous 28-day cycles
  Interventions: Drug: Tazemetostat
- Dose Escalation Level 7 (Experimental): Pediatric patients with select R/R rhabdoid tumors, INI1- SMARCA4-negative tumors, or synovial sarcoma who participated in the dose escalation portion of the study.
  Participants received 1200 mg/m^2, open-label, oral tazemetostat twice daily (BID) in continuous 28-day cycles
  Interventions: Drug: Tazemetostat
- Dose Expansion Cohort 1 (Experimental): Pediatric patients with atypical teratoid rhabdoid tumor (ATRT) who participated in the dose expansion portion of the study.
  Patients received 1200 mg/m^2 open-label, tazemetostat BID orally in continuous 28-day cycles.
  Interventions: Drug: Tazemetostat
- Dose Expansion Cohort 2 (Experimental): Pediatric patients with malignant rhabdoid tumor (MRT)/ rhabdoid tumor of kidney (RTK)/select tumors with rhabdoid features who participated in the dose expansion portion of the study
  Patients whose disease was without central nervous system (CNS) involvement received 520 mg/m^2 open-label, tazemetostat BID orally in continuous 28-day cycles. Patients whose disease had CNS involvement received 1200 mg/m^2 open-label, tazemetostat BID orally in continuous 28-day cycles.
  Interventions: Drug: Tazemetostat
- Dose Expansion Cohort 3 (Experimental): Pediatric patients with INI-negative tumors who participated in the dose expansion portion of the study.
  Patients whose disease was without central nervous system (CNS) involvement received 520 mg/m^2 open-label, tazemetostat BID orally in continuous 28-day cycles. Patients whose disease had CNS involvement received 1200 mg/m^2 open-label, tazemetostat BID orally in continuous 28-day cycles.
  Interventions: Drug: Tazemetostat
- Dose Expansion Cohort 4 (Experimental): Pediatric patients with one of the tumor types defined in Cohorts 1 through 3 or synovial sarcoma with SS18-SSX rearrangement.
  Patients received 800 mg/m^2 tazemetostat three times daily (TID) orally in continuous 28-day cycles.
  Interventions: Drug: Tazemetostat

INTERVENTIONS:
Drug: Tazemetostat — Tazemetostat (EPZ-6438) is a selective small molecule inhibitor of the histone-lysine methyltransferase EZH2 gene.
  Other Names: IPN60200; EPZ-6438; E7438

SUMMARY:
This is a Phase I, open-label, dose escalation and dose expansion study with BID (suspension) and TID (tablet) oral dose of the enhancer of zeste homolog-2 (EZH2) inhibitor, tazemetostat. Subjects will be screened for eligibility within 14 days of the planned first dose of tazemetostat. A treatment cycle will be 28 days. Response assessment will be evaluated after 8 weeks of treatment and subsequently every 8 weeks while on study.

DETAILED DESCRIPTION:
The study has two parts: Dose Escalation and Dose Expansion.

Dose escalation for subjects with the following relapsed/refractory malignancies:

* Rhabdoid tumors:
* Atypical teratoid rhabdoid tumor (ATRT)
* Malignant rhabdoid tumor (MRT)
* Rhabdoid tumor of kidney (RTK)
* Selected tumors with rhabdoid features
* Integrase interactor 1 (INI1)-negative tumors:
* Epithelioid sarcoma
* Epithelioid malignant peripheral nerve sheath tumor
* Extraskeletal myxoid chondrosarcoma
* Myoepithelial carcinoma
* Renal medullary carcinoma
* Other INI1-negative malignant tumors (e.g., dedifferentiated chordoma)
* Synovial Sarcoma with a SS18-SSX rearrangement Dose Escalation cohorts are closed to enrollment.

Dose Expansion at the maximum tolerated dose (MTD) or the recommended phase 2 dose (RP2D)

* Cohort 1 - ATRT
* Cohort 2 - MRT/RTK/selected tumors with rhabdoid features
* Cohort 3 - INI-negative tumors:
* Epithelioid sarcoma
* Epithelioid malignant peripheral nerve sheath tumor
* Extraskeletal myxoid chondrosarcoma
* Myoepithelial carcinoma
* Renal medullary carcinoma
* Chordoma (poorly differentiated or de-differentiated)
* Other INI1-negative malignant tumors (e.g., dedifferentiated chordoma)
* Cohort 4 - Tumor types eligible for Cohorts 1 through 3 or synovial sarcoma with SS18-SSX rearrangement

ELIGIBILITY:
Inclusion Criteria:

1. Age (at the time of consent/assent): ≥6 months to <18 years

   - Cohort 4 only: ≥10 years to <18 years
2. Performance Status:

   * If <12 years of age: Lanksy Performance Status >50%
   * If ≥12 years of age: Karnofsky Performance Status >50% NOTE: If subject is unable to walk due to paralysis, but is mobile in a wheelchair, subject is considered to be ambulatory for the purpose of assessing their performance status.
3. Has provided signed written informed consent/assent
4. Has a life expectancy of >3 months
5. Has relapsed or refractory disease and no standard treatment options as determined by locally or regionally available standards of care and treating physician's discretion
6. Is ineligible or inappropriate for other treatment regimens known to have effective potential
7. Has a documented local diagnostic pathology of original biopsy confirmed by a Clinical Laboratory Improvement Amendments (CLIA)/College of American Pathologists (CAP) or equivalent laboratory certification
8. Has all prior treatment (i.e., chemotherapy, immunotherapy, radiotherapy) related clinically significant toxicities resolve to ≤ Grade 1 per CTCAE, version 4.03 or are clinically stable and not clinically significant, at time of enrollment
9. Has completed a prior therapy (ies) according to the criteria below:

   * Other investigational study agent (any medicinal product that is not approved in the country of treatment for any indication, adult or pediatric) (At least 30 days or five half-lives, whichever is longer, since last dose prior to the first dose of tazemetostat)
   * Chemotherapy: cytotoxic (At least 14 days since last dose of chemotherapy prior to first dose of tazemetostat)
   * Chemotherapy: nitrosoureas (At least 6 weeks since last dose of nitrosoureas prior to first dose of tazemetostat)
   * Chemotherapy: non-cytotoxic (e.g., small molecule inhibitor) (At least 14 days since last dose of non-cytotoxic chemotherapy prior to first dose of tazemetostat)
   * Monoclonal antibody (ies) (At least 28 days since the last dose of any monoclonal antibody prior to first dose of tazemetostat)
   * Immunotherapy (e.g., tumor vaccine) At least 6 weeks since last dose of immunotherapy agent(s) prior to first dose of tazemetostat)
   * Radiotherapy (RT) (At least 14 days from last local site RT prior to first dose of tazemetostat/At least 21 days from stereotactic radiosurgery prior to first dose of tazemetostat/At least 12 weeks from craniospinal, ≥ 50% radiation of pelvis, or total body irradiation prior to first dose of tazemetostat)
   * Hematopoietic growth factor (At least 14 days from last dose of hematopoietic growth factor prior to first dose of tazemetostat)
   * Hematopoietic cell transplantation (At least 60 days from infusion of hematopoietic cells prior to first dose of tazemetostat)
10. Has adequate hematologic (bone marrow and coagulation factors), renal and hepatic function as defined by criteria below:

    * Hematologic (BM Function):

      * Hemoglobin ≥ 8 g/dL
      * Platelets ≥100,000/mm^3 (≥100 x 10^9/L)
      * ANC ≥1,000/mm^3 (≥1.0 x 10^9/L)
    * Hematologic (Coagulation Factors):

      * INR/ PTd ≤1.5 ULN
      * PTT ≤1.5 ULN
      * Fibrinogen ≥0.75 LLN
    * Renal Function (creatinine clearance or serum creatinine):

      * Calculated creatinine clearance ≥50 mL/min/1.73m^2
      * Serum creatinine 6 months to 1 year: male 0.6 mg/dL (53 µmol/L) female 0.5 mg/dL (44 µmol/L)
      * Serum creatinine 1 to < 2 years: male 0.6 mg/dL (53 µmol/L) female 0.6 mg/dL (53 µmol/L)
      * Serum creatinine 2 to < 6 years: male 0.8 mg/dL (71 µmol/L) female 0.8 mg/dL (71 µmol/L)
      * Serum creatinine 6 to <10 years: male 1 mg/dL (88 µmol/L) female 1 mg/dL (88 µmol/L)
      * Serum creatinine 10 to <13 years: male 1.2 mg/dL (106 µmol/L) female 1.2 mg/dL (106 µmol/L)
      * Serum creatinine 13 to <16 years: male 1.5 mg/dL (133 µmol/L) female 1.4 mg/dL (125 µmol/L)
      * Serum creatinine ≥16 years: male 1.7 mg/dL (150 µmol/L) female 1.4 mg/dL (125 µmol/L)
    * Hepatic Function:

      * Total bilirubin <1.5 x ULN
      * ALT or AST <3 x ULN Eligibility can be determined by either total or conjugated bilirubin
11. For subjects with CNS involvement: Subjects must have deficits that are stable for a minimum of 14 days prior to enrollment, or seizures that are stable, not increasing in frequency or severity and controlled on current anti-seizure medication(s) for a minimum of 7 days prior to enrollment NOTE: Subjects with leptomeningeal disease or brain tumors with positive cerebral spinal fluid cytology are eligible for this study. Subjects may receive glucocorticoids (at stable or tapering dose) to control CNS symptoms prior to enrollment; however, subjects should receive a stable or tapering dose for at least 7 days prior to enrollment.
12. Has a shortening fraction of >27% or an ejection fraction of ≥50% by echocardiogram or multi-gated acquisition scan and New York Heart Association Class<2
13. Has a QT interval corrected by Fridericia's formula (QTcF) ≤450 msec
14. Is able to swallow and retain orally administered medication and does not have any uncontrolled gastrointestinal (GI) condition such as nausea, vomiting, or diarrhea, or any clinically significant GI abnormalities that may alter absorption such as malabsorption syndromes, hereditary fructose intolerance, glucose-galactose malabsorption, sucrose-isomaltase insufficiency, or major resection of stomach and/or bowels NOTE: Nasogastric and gastrostomy tube administration of the oral suspension formulation of study drug is permitted.
15. Has sufficient tumor tissue (slides or blocks) available for central confirmatory testing of immunohistochemistry and/or cytogenetics/fluorescence in situ hybridization (FISH) and/or deoxyribonucleic acid mutation analysis (required for study entry but enrollment based on local results)
16. Is willing and able to comply with all aspects of the protocol as judged by Investigator
17. For female subjects of childbearing potential: Subject must:

    * Have a negative beta-human chorionic gonadotropin (β-hCG) pregnancy test at time of Screening and within 72 hours prior to planned first dose of tazemetostat (urine or serum test is acceptable however, positive urine tests must be confirmed with serum testing), and
    * Agree to use effective contraception, as defined in Section 8.6.11 start of Screening until 6 months following the last dose of study treatment and have a male partner who uses a condom, or
    * Practice true abstinence (when this is in line with the preferred and usual lifestyle of the subject, see Section 8.6.11, or
    * Have a male partner who is vasectomized with confirmed azoospermia
18. For male subjects with a female partner of childbearing potential: Subject must:

    * Be vasectomized or
    * Agree to use condoms as defined in Section 8.5.11 from first dose of tazemetostat until 3 months following the last dose of tazemetostat, or
    * Have a female partner who is NOT of childbearing potential

For Dose Escalation Only:

To be eligible for enrollment in dose escalation, a subject must meet ALL of the following criteria in addition to the inclusion criteria listed above for all subjects:

1. Has evaluable disease as defined as lesions that can be accurately measured at least in one dimension by radiographic examination or physical examination and other lesions such as bone lesions, leptomeningeal disease, ascites, hepatosplenomegaly from disease.
2. Has one of the following histologically confirmed tumors: (NOTE: Evidence of diagnostic pathology of original biopsy confirmed by a CLIA/CAP certified laboratory must be available)

   * Rhabdoid tumor:

     * ATRT
     * MRT
     * RTK
     * Selected tumors with rhabdoid features
   * NI1-negative tumor:

     * Epithelioid sarcoma
     * Epithelioid malignant peripheral nerve sheath tumor
     * Extraskeletal myxoid chondrosarcoma
     * Myoepithelial carcinoma
     * Renal medullary carcinoma
     * Other INI1-negative malignant tumors (e.g., dedifferentiated chordoma) with Sponsor approval
   * Synovial sarcoma with SS18-SSX rearrangement (NOTE: Evidence of diagnostic pathology of original biopsy confirmed by a CLIA/CAP certified laboratory must be available) (Closed to enrollment)
3. For subjects with ATRT, MRT, RTK, or selected tumors with rhabdoid features only: the following test results must be available: Morphology and immunophenotypic panel consistent with rhabdoid tumor and Loss of INI1 or SMARCA4 confirmed by IHC, or Molecular confirmation of tumor bi-allelic INI1 or SMARCA4 loss/mutation when INI1 or SMARCA4 IHC is equivocal or unavailable
4. For subjects with INI1 negative tumor only:

   the following test results must be available: Morphology and immunophenotypic panel consistent with INI1-negative tumors, and Loss of INI1 confirmed by IHC, or Molecular confirmation of tumor bi-allelic INI1 loss/mutation when INI1 IHC is equivocal or unavailable
5. For subjects with synovial sarcoma only:

The following test results must be available:

Morphology consistent with synovial sarcoma, and Cytogenetics or FISH and/or molecular confirmation (e.g., DNA sequencing) of SS18 rearrangement t(X;18)(p11;q11)

For Dose Expansion Only:

Note: To be eligible for enrollment in Dose Expansion, a subject must meet ALL of the following criteria in addition to the inclusion criteria for ALL subjects listed above

1. Has measurable disease
2. Has one of the following histologically confirmed tumors:

   * Cohort 1 - ATRT (Closed to enrollment)
   * Cohort 2 - MRT/RTK/selected tumors with rhabdoid features (Closed to enrollment)
   * Cohort 3 - INI-negative tumors (Closed to enrollment):

     * Epithelioid sarcoma
     * Epithelioid malignant peripheral nerve sheath tumor
     * Extraskeletal myxoid chondrosarcoma(EMC)
     * Myoepithelial carcinoma
     * Renal medullary carcinoma
     * Chordoma (poorly differentiated or de-differentiated)
     * Other INI1-negative malignant tumors (e.g., dedifferentiated chordoma) with Sponsor approval
   * Cohort 4 - Tumor types eligible for Cohorts 1 through 3 or synovial sarcoma with SS18-SSX rearrangement (Closed to enrollment) NOTE: Evidence of diagnostic pathology of original biopsy confirmed by a CLIA/CAP or other Sponsor-approved certified laboratory must be available.
3. For subjects with ATRT/MRT/RTK only - have the following test results available:

   * Morphology and immunophenotypic panel consistent with rhabdoid tumor, and
   * Loss of INI1 or SMARCA4 confirmed by IHC, or
   * Molecular confirmation of tumor bi-allelic INI1 or SMARCA4 loss/mutation when INI1 or SMARCA4 IHC is equivocal or unavailable
4. For subjects with INI1-negative tumors only: The following test results must be available:

   * Morphology and immunophenotypic panel consistent with INI1-negative tumors, and
   * Loss of INI1 confirmed by IHC, or
   * Molecular confirmation of tumor bi-allelic INI1 loss/mutation when INI1 IHC is equivocal or unavailable
5. For subjects with synovial sarcoma with SS18-SSX rearrangement (in Cohort 4 ONLY - Closed to enrollment): The following test results must be available:

   * Morphology consistent with synovial sarcoma, and
   * Cytogenetics or FISH and/or molecular confirmation (e.g., deoxyribonucleic acid [DNA] sequencing) of SS18 rearrangement t(X;18)(p11;q11)
6. For subjects to be enrolled in Cohort 4 (Closed to enrollment): Able to swallow and retain orally administered tablets

Exclusion Criteria:

1. Has had prior exposure to tazemetostat or other inhibitor(s) of EZH2
2. Is being actively treated for another concurrent malignancy or is less than five years from completion of treatment for another malignancy
3. Has participated in another interventional clinical study and received investigational drug within 30 days or 5 half-lives, whichever is longer, prior to the planned first dose of tazemetostat
4. Has had major surgery within 2 weeks prior to enrollment NOTE: Minor surgery (e.g., minor biopsy of extracranial site, central venous catheter placement, shunt revision) is permitted within 2 weeks prior to enrollment.
5. Has thrombocytopenia, neutropenia, or anemia of Grade ≥3 (per CTCAE 4.03 criteria) or any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS). Has abnormalities known to be associated with MDS (e.g. del 5q, chr 7 abn) and MPN (e.g. JAK2 V617F) observed in cytogenetic testing and DNA sequencing.

   Note: Bone marrow aspirate/biopsy will be conducted following abnormal peripheral blood smear morphology assessment conducted by central lab at screening. Cytogenetic testing and DNA sequencing will be conducted following an abnormal result of bone marrow aspirate/biopsy.
6. Has a prior history of T-LBL/T-ALL.
7. Has clinically active heart disease including prolonged corrected QTcF (>450 msec)
8. Is currently taking any prohibited medication(s) as described in Section 7.3.
9. Is unwilling to exclude grapefruit juice, Seville oranges and grapefruit from the diet and all foods that contain those fruits from time of enrollment to while on study
10. Has an active infection requiring systemic treatment
11. Is immunocompromised (i.e. congenital immunodeficiencies), including subjects known history of infection with human immunodeficiency virus (HIV)
12. Has known history of chronic infection with hepatitis B virus (hepatitis B surface antigen positive) or hepatitis C virus (detectable HCV RNA)
13. Has had a symptomatic venous thrombosis within the 14 days prior to study enrollment NOTE: Subjects with a history of a deep vein thrombosis 14 days prior to study enrollment who are on anticoagulation therapy with low molecular weight heparin are eligible for this study
14. For subjects with CNS involvement (primary tumor or metastatic disease): Have any active bleeding, or new intratumoral hemorrhage of more than punctate size on Screening MRI obtained within 14 days of starting study drug,or known bleeding diathesis or treatment with anti-platelet or anti-thrombotic agents 15.15. Has known hypersensitivity to any of the components of tazemetostat or other inhibitor(s) of EZH2, or hypersensitivity to Ora-sweet or methylparaben

16. Has an uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, or psychiatric illness/social situations that would limit compliance with study requirements 17. For female subjects of childbearing potential: Is pregnant or nursing For male subjects: Is unwilling to adhere to contraception criteria from time of enrollment in study to at least 30 days after last dose of tazemetostat.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2021-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical, Study Director — Ipsen
Locations (35):
- United States (17):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California San Francisco - Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - John Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital - Cancer Center, Boston, Massachusetts
  - Memorial Sloan Kettering, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Inc., Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Children's Cancer and Hematology Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (4):
  - Sydney Children's Hospital, Sydney, New South Wales
  - Lady Cilento/Queensland Children's Hospital, South Brisbane, Queensland
  - The Royal Children's Hospital, Melbourne, Victoria
  - The Childrens Hospital at Westmead Oncology Unit, Westmead
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Rigshospitalet Department of Oncology Blegdamsvej, Copenhagen, Denmark
- France (2):
  - Institut Curie, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Children's Hospital Augsburg Klinikum, Augsburg
  - Charite - Universitatsmedizin Berlin, Berlin
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Westfalische Wilhelms - Universitat Munster Padiatrische, Münster
- Italy (2):
  - Istituto Giannina Gaslini- UOSD Centro di Neuro-Oncologia, Genova
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
- Netherlands (2):
  - Erasmus University Medical Center - Sophia Children's Hospital, Rotterdam
  - Prinses Maxima Centrum voor Kinderoncologie, Utrecht
- United Kingdom (2):
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Central Manchester University Hospital - Royal Manchester Children's Hospital, Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Escalation Level 1: Patients with relapsed/refractory rhabdoid tumors, integrase interactor 1 (INI1)-negative tumors, or synovial sarcoma with SS18-SSX rearrangement received oral tazemetostat 240 milligrams per square meter (mg/m^2) twice daily (BID) in continuous 28-day cycles.
- Dose Escalation Level 2: Patients with relapsed/refractory rhabdoid tumors, INI1-negative tumors, or synovial sarcoma with SS18-SSX rearrangement received oral tazemetostat 300 mg/m^2 BID in continuous 28-day cycles.
- Dose Escalation Level 3: Patients with relapsed/refractory rhabdoid tumors, INI1-negative tumors, or synovial sarcoma with SS18-SSX rearrangement received oral tazemetostat 400 mg/m^2 BID in continuous 28-day cycles.
- Dose Escalation Level 4: Patients with relapsed/refractory rhabdoid tumors, INI1-negative tumors, or synovial sarcoma with SS18-SSX rearrangement received oral tazemetostat 520 mg/m^2 BID in continuous 28-day cycles.
- Dose Escalation Level 5: Patients with relapsed/refractory rhabdoid tumors, INI1-negative tumors, or synovial sarcoma with SS18-SSX rearrangement received oral tazemetostat 700 mg/m^2 BID in continuous 28-day cycles.
- Dose Escalation Level 6: Patients with relapsed/refractory rhabdoid tumors, INI1-negative tumors, or synovial sarcoma with SS18-SSX rearrangement received oral tazemetostat 900 mg/m^2 BID in continuous 28-day cycles.
- Dose Escalation Level 7: Patients with relapsed/refractory rhabdoid tumors, INI1-negative tumors, or synovial sarcoma with SS18-SSX rearrangement received oral tazemetostat 1200 mg/m^2 BID in continuous 28-day cycles.
- Dose Expansion Cohort 1: Patients with atypical teratoid rhabdoid tumor (ATRT) who participated in the dose expansion portion of the study received 1200 mg/m^2 open-label, tazemetostat BID orally in continuous 28-day cycles.
- Dose Expansion Cohort 2: Patients with malignant rhabdoid tumor (MRT)/ rhabdoid tumor of kidney (RTK)/select tumors with rhabdoid features who participated in the dose expansion portion of the study. Patients whose disease was without central nervous system (CNS) involvement received 520 mg/m^2 open-label, tazemetostat BID orally in continuous 28-day cycles. Patients whose disease had CNS involvement received 1200 mg/m^2 open-label, tazemetostat BID orally in continuous 28-day cycles.
- Dose Expansion Cohort 3: Patients with INI-negative tumors who participated in the dose expansion portion of the study. Patients whose disease was without central nervous system (CNS) involvement received 520 mg/m^2 open-label, tazemetostat BID orally in continuous 28-day cycles. Patients whose disease had CNS involvement received 1200 mg/m^2 open-label, tazemetostat BID orally in continuous 28-day cycles.
- Dose Expansion Cohort 4: Patients with one of the tumor types defined in Cohorts 1 through 3 or synovial sarcoma with SS18-SSX rearrangement received 800 mg/m^2 tazemetostat three times daily (TID) orally in continuous 28-day cycles.
Period: Period 1: Dose Escalation Phase
Arm/Group | Dose Escalation Level 1 | Dose Escalation Level 2 | Dose Escalation Level 3 | Dose Escalation Level 4 | Dose Escalation Level 5 | Dose Escalation Level 6 | Dose Escalation Level 7 | Dose Expansion Cohort 1 | Dose Expansion Cohort 2 | Dose Expansion Cohort 3 | Dose Expansion Cohort 4
Started | 8 | 6 | 6 | 7 | 6 | 6 | 7 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 6 | 6 | 6 | 6 | 5 | 7 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Patient refused further treatment of study drug | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Unacceptable toxicity | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 7 | 6 | 5 | 6 | 6 | 4 | 6 | 0 | 0 | 0 | 0
Period: Period 2: Dose Expansion Cohort
Arm/Group | Dose Escalation Level 1 | Dose Escalation Level 2 | Dose Escalation Level 3 | Dose Escalation Level 4 | Dose Escalation Level 5 | Dose Escalation Level 6 | Dose Escalation Level 7 | Dose Expansion Cohort 1 | Dose Expansion Cohort 2 | Dose Expansion Cohort 3 | Dose Expansion Cohort 4
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 20 | 18 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 20 | 18 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Patient refused further treatment of study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 17 | 14 | 4
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all patients who received at least one dose of tazemetostat.
Groups:
- Dose Escalation Level 1: Patients with relapsed/refractory rhabdoid tumors, INI1-negative tumors, or synovial sarcoma with SS18-SSX rearrangement received oral tazemetostat 240 mg/m^2 BID in continuous 28-day cycles.
- Dose Expansion Cohort 1: Patients with ATRT who participated in the dose expansion portion of the study received 1200 mg/m^2 open-label, tazemetostat BID orally in continuous 28-day cycles.
- Dose Expansion Cohort 2: Patients with MRT/ RTK/select tumors with rhabdoid features who participated in the dose expansion portion of the study. Patients whose disease was without CNS involvement received 520 mg/m^2 open-label, tazemetostat BID orally in continuous 28-day cycles. Patients whose disease had CNS involvement received 1200 mg/m^2 open-label, tazemetostat BID orally in continuous 28-day cycles.
- Dose Expansion Cohort 3: Patients with INI-negative tumors who participated in the dose expansion portion of the study.
  Patients whose disease was without CNS involvement received 520 mg/m^2 open-label, tazemetostat BID orally in continuous 28-day cycles. Patients whose disease had CNS involvement received 1200 mg/m^2 open-label, tazemetostat BID orally in continuous 28-day cycles.
- Dose Expansion Cohort 4: Patients with one of the tumor types defined in Cohorts 1 through 3 or synovial sarcoma with SS18-SSX rearrangement received 800 mg/m^2 tazemetostat TID orally in continuous 28-day cycles.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Level 1 | Dose Escalation Level 2 | Dose Escalation Level 3 | Dose Escalation Level 4 | Dose Escalation Level 5 | Dose Escalation Level 6 | Dose Escalation Level 7 | Dose Expansion Cohort 1 | Dose Expansion Cohort 2 | Dose Expansion Cohort 3 | Dose Expansion Cohort 4 | Total
Number analyzed (Participants) | 8 | 6 | 6 | 7 | 6 | 6 | 7 | 19 | 20 | 18 | 6 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 6 | 6 | 7 | 6 | 6 | 7 | 19 | 20 | 17 | 4 | 106
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.5 (1.89) | 11.5 (5.24) | 4.6 (3.98) | 4.5 (3.50) | 7.0 (4.82) | 4.0 (2.79) | 4.8 (4.97) | 4.4 (4.25) | 3.4 (3.31) | 12.8 (5.26) | 14.7 (3.61) | 6.6 (5.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 5 | 2 | 4 | 2 | 12 | 7 | 11 | 3 | 59
  Male | 4 | 2 | 1 | 2 | 4 | 2 | 5 | 7 | 13 | 7 | 3 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 5 | 2 | 4 | 1 | 17
  Not Hispanic or Latino | 8 | 4 | 2 | 7 | 4 | 5 | 5 | 13 | 14 | 12 | 5 | 79
  Unknown or Not Reported | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 1 | 4 | 2 | 0 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 8
  White | 7 | 6 | 4 | 5 | 4 | 4 | 5 | 14 | 12 | 14 | 4 | 79
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 7 | 3 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) (Dose Escalation Only)
Description: The incidence and severity of treatment-emergent adverse events qualifying as protocol-defined dose-limiting toxicities that occurred during the first month of treatment was used to determine the RP2D and/or maximum tolerated dose (MTD) in pediatric patients treated with tazemetostat.
Time Frame: Cycle 1, from the start of study treatment (Day 1) until the end of the first Cycle (Day 28) of treatment
Population: The ITT population included all patients who received at least one dose of tazemetostat.
Measure: Number; unit: mg/m^2 BID
Groups:
- Overall Dose Escalation: Patients with relapsed/refractory rhabdoid tumors, INI1-negative tumors, or synovial sarcoma with SS18-SSX rearrangement received oral tazemetostat at BID dose level 1: 240 mg/m^2, dose level 2: 300 mg/m^2, dose level 3: 400 mg/m^2, dose level 4: 520 mg/m^2, dose level 5: 700 mg/m^2, dose level 6: 900 mg/m^2 and dose level 7: 1200 mg/m^2 in continuous 28-day cycles.
Arm/Group | Overall Dose Escalation
Number analyzed (Participants) | 46
mg/m^2 BID
  RP2D for patients with ATRT or CNS involvement | 1200
  RP2D for patients without CNS involvement | 520

2. Primary Outcome: Number of Dose-limiting Toxicities (Dose Escalation Only)
Description: The RP2D in pediatric patients treated with tazemetostat as determined by the incidence and severity of treatment-emergent adverse events qualifying as protocol-defined dose-limiting toxicities that occurred during the first month of treatment.
Time Frame: Cycle 1, from the start of study treatment (Day 1) until the end of the first Cycle (Day 28) of treatment
Population: Dose-Limiting Toxicity (DLT) population included all patients in the safety population set who experienced a DLT during Cycle 1 or were not removed from Cycle 1 for reasons other than toxicity and did not have an interruption in study treatment for more than 14 days during Cycle 1. Only those patients with data collected at Cycle 1 are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Level 1 | Dose Escalation Level 2 | Dose Escalation Level 3 | Dose Escalation Level 4 | Dose Escalation Level 5 | Dose Escalation Level 6 | Dose Escalation Level 7
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 1 | 0 | 0 | 0 | 1 | 0

3. Primary Outcome: Overall Response Rate (ORR) (Dose Expansion Only)
Description: ORR is defined as the percentage of patients who achieved a confirmed complete response (CR) and/or partial response (PR) defined by response evaluation criteria in solid tumors (RECIST) or response assessment in neuro-oncology (RANO) criteria from the start of tazemetostat treatment until disease progression or the start of subsequent anticancer therapy, whichever occurs first. CR is defined as disappearance of all target and non-target lesions (with all lymph nodes must be non-pathological in size or under 10 millimeters [mm] in short axis) and PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR= CR+PR.
Time Frame: RECIST assessments performed at screening (within 14 days before start of study intervention) and every 8 weeks post start of dosing, approximately up to 302 weeks
Population: The ITT population included all patients who received at least one dose of tazemetostat.
Measure: Number; unit: Percentage of participants
Arm/Group | Dose Expansion Cohort 1 | Dose Expansion Cohort 2 | Dose Expansion Cohort 3 | Dose Expansion Cohort 4
Number analyzed (Participants) | 19 | 20 | 18 | 6
Percentage of participants | 26.3 | 0 | 16.7 | 16.7

4. Secondary Outcome: ORR (Dose Escalation Only)
Description: ORR is defined as the percentage of patients who achieved a confirmed CR and/or PR defined by RECIST or RANO criteria from the start of tazemetostat treatment until disease progression or the start of subsequent anticancer therapy, whichever occurs first. CR is defined as disappearance of all target and non-target lesions (with all lymph nodes must be non-pathological in size or under 10 mm in short axis) and PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR= CR+PR.
Time Frame: as for outcome 3
Population: The ITT population included all patients who received at least one dose of tazemetostat.
Measure: Number; unit: Percentage of participants
Arm/Group | Dose Escalation Level 1 | Dose Escalation Level 2 | Dose Escalation Level 3 | Dose Escalation Level 4 | Dose Escalation Level 5 | Dose Escalation Level 6 | Dose Escalation Level 7
Number analyzed (Participants) | 8 | 6 | 6 | 7 | 6 | 6 | 7
Percentage of participants | 0 | 0 | 0 | 14.3 | 16.7 | 16.7 | 0

5. Secondary Outcome: Progression Free Survival (PFS) (Dose Expansion Only)
Description: PFS was defined as the interval of time (in weeks) from the date of first dose of study drug and the earliest date of disease progression or death, from any cause defined by RECIST or RANO criteria. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (including at least a 5 mm absolute increase). The presence of new lesions also constitutes to disease progression.
Time Frame: as for outcome 3
Population: The ITT population included all patients who received at least one dose of tazemetostat.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dose Expansion Cohort 1 | Dose Expansion Cohort 2 | Dose Expansion Cohort 3 | Dose Expansion Cohort 4
Number analyzed (Participants) | 19 | 20 | 18 | 6
weeks | 7.9 [6.0 to 24.3] | 7.7 [3.4 to 8.0] | 15.9 [8.0 to 21.3] | 28.3 [7.9 to 145.4]

6. Secondary Outcome: Overall Survival (Dose Expansion Only)
Description: Overall survival was defined as the time (in weeks) from the first dose of study drug to the date of death due to any cause.
Time Frame: as for outcome 3
Population: The ITT population included all patients who received at least one dose of tazemetostat.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dose Expansion Cohort 1 | Dose Expansion Cohort 2 | Dose Expansion Cohort 3 | Dose Expansion Cohort 4
Number analyzed (Participants) | 19 | 20 | 18 | 6
weeks | 21.4 [11.0 to 50.3] | 14.1 [6.9 to 22.4] | 41.8 [18.6 to 55.6] | 103.1 [12.3 to 185.6]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the time of the first dose of study treatment (Day 1) until the earlier of either 30 days after the discontinuation of study treatment or until the initiation of subsequent anticancer therapy, approximately 114 weeks (dose escalation phase) and 138.7 weeks (dose expansion phase). All-cause mortality (deaths) were collected from the time of the first dose of study treatment (Day 1) up to 302 weeks.
Description: The safety population consists of all patients in the ITT population who had at least one post-dose safety observation recorded.
Arm/Group | Dose Escalation Level 1 | Dose Escalation Level 2 | Dose Escalation Level 3 | Dose Escalation Level 4 | Dose Escalation Level 5 | Dose Escalation Level 6 | Dose Escalation Level 7 | Dose Expansion Cohort 1 | Dose Expansion Cohort 2 | Dose Expansion Cohort 3 | Dose Expansion Cohort 4
All-Cause Mortality (participants affected / at risk) | 7/8 | 6/6 | 4/6 | 4/7 | 5/6 | 4/6 | 7/7 | 15/19 | 18/20 | 16/18 | 4/6
Serious Adverse Events (participants affected / at risk) | 4/8 | 1/6 | 3/6 | 2/7 | 3/6 | 4/6 | 2/7 | 12/19 | 10/20 | 9/18 | 3/6
Other Adverse Events (participants affected / at risk) | 8/8 | 5/6 | 6/6 | 7/7 | 6/6 | 6/6 | 6/7 | 19/19 | 19/20 | 18/18 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Dose Escalation Level 1 (N=8) | Dose Escalation Level 2 (N=6) | Dose Escalation Level 3 (N=6) | Dose Escalation Level 4 (N=7) | Dose Escalation Level 5 (N=6) | Dose Escalation Level 6 (N=6) | Dose Escalation Level 7 (N=7) | Dose Expansion Cohort 1 (N=19) | Dose Expansion Cohort 2 (N=20) | Dose Expansion Cohort 3 (N=18) | Dose Expansion Cohort 4 (N=6)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (7) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Central Nervous System Ventriculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mastoid abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulval abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/11 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Unintentional medical device removal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhabdoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 1 (2)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Level 1 (N=8) | Dose Escalation Level 2 (N=6) | Dose Escalation Level 3 (N=6) | Dose Escalation Level 4 (N=7) | Dose Escalation Level 5 (N=6) | Dose Escalation Level 6 (N=6) | Dose Escalation Level 7 (N=7) | Dose Expansion Cohort 1 (N=19) | Dose Expansion Cohort 2 (N=20) | Dose Expansion Cohort 3 (N=18) | Dose Expansion Cohort 4 (N=6)
Otitis media (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (9) | 1 (1) | 1 (2) | 1 (1) | 2 (3) | 1 (1) | 3 (3) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (4) | 2 (2) | 1 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 1 (4) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 3 (3) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (3) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 1 (3) | 2 (4) | 4 (29) | 8 (18) | 5 (13) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (7)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (2) | 0 (0) | 1 (1) | 5 (5) | 4 (4) | 4 (4) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 2 (2) | 0 (0) | 1 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 1 (1) | 2 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 2 (3) | 2 (2) | 1 (2) | 4 (6) | 1 (1) | 7 (9) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Paraesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (2)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (3) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 3 (5) | 3 (9) | 2 (2) | 6 (11) | 4 (5) | 6 (8) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (3) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (3) | 3 (5) | 2 (4) | 3 (7) | 2 (4) | 6 (12) | 11 (19) | 9 (14) | 11 (34) | 5 (19)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (6) | 1 (1) | 3 (5) | 2 (3) | 1 (1) | 6 (6) | 5 (5) | 11 (16) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 2 (3) | 4 (6) | 2 (6) | 1 (1) | 7 (12) | 3 (3) | 7 (11) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (4) | 1 (2) | 0 (0) | 1 (1) | 4 (4) | 3 (6) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (5) | 2 (4) | 1 (1) | 4 (6) | 5 (8) | 7 (16) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 2 (3) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 4 (4) | 2 (2) | 5 (7) | 2 (3)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 5 (6) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (11) | 1 (1) | 3 (3)
Lymphocyte count decreased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 3 (3) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (8)
Blood bromide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (5) | 0 (0) | 3 (6) | 0 (0) | 1 (4) | 2 (7) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Behaviour disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fear (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmetria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Auditory nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IIIrd nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IVth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuromyopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIth nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Defect conduction intraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth development disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site erosion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | 1 (2)
Weight increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corneal epithelium defect (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exophthalmos (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gaze palsy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurotrophic keratopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deafness transitory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal rash (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT02601937/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT02601937/SAP_001.pdf